CLINICAL TRIAL: NCT02833948
Title: Randomized Comparison of a Rivaroxaban-based Strategy With an Antiplatelet-based Strategy Following Successful TAVR for the Prevention of Leaflet Thickening and Reduced Leaflet Motion as Evaluated by Four-dimensional, Volume-rendered Computed Tomography (4DCT) - Substudy of the GALILEO-trial
Brief Title: Comparison of a Rivaroxaban-based Strategy With an Antiplatelet-based Strategy Following Successful TAVR for the Prevention of Leaflet Thickening and Reduced Leaflet Motion as Evaluated by Four-dimensional, Volume-rendered Computed Tomography (4DCT)
Acronym: GALILEO-4D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ECRI bv (Industry)
Collaborators: Rigshospitalet, Denmark (Other); Bayer (Industry); Cardialysis BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ECRI 006 - H-15016807
Record Dates: First submitted 2016-06-24; First posted 2016-07-14 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Aortic Valve Stenosis; Cardiovascular Diseases; Heart Valve Diseases; Ventricular Outflow Obstruction; Thrombosis
Keywords: Heart Valve Disease; Randomized Controlled Trial; Transcatheter Aortic Valve Replacement; TAVR; Valve Thrombosis
MeSH Terms: conditions — Aortic Valve Stenosis; Cardiovascular Diseases; Heart Valve Diseases; Ventricular Outflow Obstruction; Thrombosis | interventions — Aspirin; acetylsalicylic acid lysinate; Clopidogrel; Rivaroxaban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ASA + Clopidogrel (Active Comparator): ASA (Acetylsalicylic acid) 75-100mg + Clopidogrel 75mg for 90 days, followed by ASA 75-100mg monotherapy
  Interventions: Drug: Acetylsalicylic acid; Drug: Clopidogrel
- Rivaroxaban + ASA (Experimental): Rivaroxaban 10mg + ASA 75-100mg for 90 days, followed by rivaroxaban 10mg monotherapy
  Interventions: Drug: Acetylsalicylic acid; Drug: Rivaroxaban

INTERVENTIONS:
Drug: Acetylsalicylic acid — Drug: Acetylsalicylic acid:
  75 - 100 mg OD (for first 90 days only in arm 1)
  Other Names: Asprin
Drug: Clopidogrel — Drug: Clopidogrel 75 mg OD for first 90 days
  Other Names: Plavix
  Arms: ASA + Clopidogrel
Drug: Rivaroxaban — Drug: Rivaroxaban (Xarelto):
  10 mg OD (once-daily)
  Other Names: Xarelto
  Arms: Rivaroxaban + ASA

SUMMARY:
The aortic valve is located between the left ventricle and the aorta. Patients with symptomatic, severe aortic valve stenosis conventionally have it surgically replaced requiring direct access to the heart through the chest. Transcatheter aortic valve replacement (TAVR) is now a well-established alternative for treating severe aortic valve stenosis. Both types of intervention improve prognosis and alleviate symptoms.

The optimal choice of blood thinning therapy after TAVR is unknown. It has been reported that leaflet thrombosis with reduced leaflet motion can occur and this phenomenon has been suggested to be potentially related with neurological events. In addition, the occurence of this phenomenon can be reduced with anticoagulation blood thinning therapy.

The purpose of this study is to evaluate if anticoagulation compared to the usual double platelet inhibitor therapy after TAVR can reduce the risk of leaflet thrombosis.

DETAILED DESCRIPTION:
BACKGROUND: Transcatheter aortic valve replacement (TAVR) has become an established therapeutic option for patients with symptomatic, severe aortic valve stenosis, who are ineligible or at high risk for conventional surgical aortic valve replacement (SAVR). It was recently reported that leaflet thickening and reduced leaflet motion, verified by four-dimensional computed tomography (4DCT), was not uncommon after both TAVR and SAVR. It has been emphasized that this phenomenon should be further investigated for its effect on clinical outcomes (e.g. stroke) and valve durability. As this valve leaflet thickening and reduced motion could be reversed by oral anticoagulant (OAC) treatment and was not observed in patients on chronic OAC therapy, it has been hypothesized that this phenomenon could be related to possible leaflet thrombosis or a "thrombotic film" on the leaflets.

AIM: To evaluate whether a rivaroxaban-based strategy, following successful TAVR, compared to an antiplatelet-based strategy, is superior in reducing subclinical valve leaflet thickening and motion abnormalities - as detected by 4DCT-scan.

POPULATION: All patients undergoing successful TAVR by ileofemoral or subclavian access with an approved TAVR device will be screened for eligibility. Included subjects must provide written informed consent. Inclusion and exclusion criteria are listed below.

DESIGN: The GALILEO-4D trial will be conducted as a substudy of the multicenter, open-label, randomized, event-driven, active-controlled GALILEO trial. Patients will be 1:1 randomized to an antiplatelet-based strategy vs. rivaroxaban-based strategy - the randomization will adopt the same 1:1 randomization of the main GALILEO trial. In case the GALILEO-4D trial should still be continued after completion of the main GALILEO trial, this 1:1 randomization will be continued until inclusion of 150 patients in both treatment groups. In total, 300 patients will be randomized in the GALILEO-4D trial.

INTERVENTION: Subjects in the GALILEO-4D substudy will receive the same intervention as in the main GALILEO study. In addition, a 4DCT-scan and echocardiography will be performed at 90 days after randomization.

END POINTS: The primary endpoint constitutes the rate of patients with at least one prosthetic leaflet with > 50% motion reduction as assessed by cardiac 4DCT-scan (total N = 300). The secondary endpoints are listed below.

ELIGIBILITY:
Inclusion Criteria:

* Successful TAVR of a native aortic valve stenosis
* By iliofemoral or subclavian access
* With any approved/marketed TAVR device
* Written informed consent

Exclusion Criteria:

* Atrial fibrillation (AF), current or previous, with an ongoing indication for oral anticoagulant treatment
* Any other indication for continued treatment with any oral anticoagulant
* Known bleeding diathesis (such as but not limited to platelet count ≤ 50,000/mm3 at screening, hemoglobin level < 8.5 g/dL or < 5.3 mmol/l, history of intracranial hemorrhage, or subdural hematoma)
* Any indication for dual antiplatelet therapy (DAPT) for more than three months after randomization (such as coronary, carotid, or peripheral stent implantation)
* Clinically overt stroke within the last three months
* Planned coronary or vascular intervention or major surgery
* Severe renal insufficiency (eGFR < 30 mL/min/1.73 m2) or on dialysis, or post-TAVR unresolved acute kidney injury with renal dysfunction ≥ stage 2
* Moderate and severe hepatic impairment (Child-Pugh Class B or C) or any hepatic disease associated with coagulopathy
* Iodine contrast allergy or other condition that prohibits CT imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2016-05; Primary Completion 2018-12 (Actual); Study Completion 2019-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Søndergaard, MD;DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (25):
- United States (4):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mount Sinai M.C, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas, Health Science Center, Houston, Texas
- Canada (2):
  - University of Alberta Hospital, Edmonton
  - Providence Health Care, Vancouver
- Denmark (3):
  - Aarhus university hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- Germany (9):
  - Kerckhoff Klinik GmbH, Bad Nauheim
  - Charité- Universitätsmedizin Berlin - Campus Mitte, Berlin
  - Deutsches Herzzentrum Berlin, Berlin
  - St. Johannes Hospital, Dortmund
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Medicin Herzzentrum Lahr/Baden, Lahr
  - Herzzentrum Leipzig - Universitätsklinik, Leipzig
  - Deutsches Herzzentrum München, München
- Netherlands (3):
  - Academic Medical Center, Amsterdam
  - Amphia Zienkenhuis, Breda
  - Erasmus M.C, Rotterdam
- Sweden (2):
  - Skåne University Hospital, Lund
  - Karolinska University Hospital, Stockholm
- Switzerland (2):
  - University Hospital Basel, Basel
  - Inselspital, Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makkar RR, Fontana G, Jilaihawi H, Chakravarty T, Kofoed KF, De Backer O, Asch FM, Ruiz CE, Olsen NT, Trento A, Friedman J, Berman D, Cheng W, Kashif M, Jelnin V, Kliger CA, Guo H, Pichard AD, Weissman NJ, Kapadia S, Manasse E, Bhatt DL, Leon MB, Sondergaard L. Possible Subclinical Leaflet Thrombosis in Bioprosthetic Aortic Valves. N Engl J Med. 2015 Nov 19;373(21):2015-24. doi: 10.1056/NEJMoa1509233. Epub 2015 Oct 5. PMID 26436963
- [Derived] De Backer O, Dangas GD, Jilaihawi H, Leipsic JA, Terkelsen CJ, Makkar R, Kini AS, Veien KT, Abdel-Wahab M, Kim WK, Balan P, Van Mieghem N, Mathiassen ON, Jeger RV, Arnold M, Mehran R, Guimaraes AHC, Norgaard BL, Kofoed KF, Blanke P, Windecker S, Sondergaard L; GALILEO-4D Investigators. Reduced Leaflet Motion after Transcatheter Aortic-Valve Replacement. N Engl J Med. 2020 Jan 9;382(2):130-139. doi: 10.1056/NEJMoa1911426. Epub 2019 Nov 16. PMID 31733182

RESULTS

PARTICIPANT FLOW:
Groups:
- ASA + Clopidogrel: ASA (Acetylsalicylic acid) 75-100mg + Clopidogrel 75mg for 90 days, followed by ASA 75-100mg monotherapy
  Acetylsalicylic acid: Drug: Acetylsalicylic acid:
  75 - 100 mg OD (for first 90 days only in arm 1)
  Clopidogrel: Drug: Clopidogrel 75 mg OD for first 90 days
  If new-onset atrial fibrillation occurred within three months, clopidogrel was replaced by vitamin K antagonist targeting an international normalized ratio of 2 to 3 and combined with acetylsalicyclic acid 75mg to 100mg once-daily (which was discontinued at three month post-TAVR); however, if new-onset atrial fibrillation occurred after three months, acetylsalicyclic acid 75mg to 100mg once-daily was replaced by vitamin K antagonist targeting an international normalized ratio of 2 to 3.
- Rivaroxaban + ASA: Rivaroxaban 10mg + ASA 75-100mg for 90 days, followed by rivaroxaban 10mg monotherapy
  Acetylsalicylic acid: Drug: Acetylsalicylic acid:
  75 - 100 mg OD (for first 90 days only in arm 1)
  Rivaroxaban: Drug: Rivaroxaban (Xarelto):
  10 mg OD (once-daily)
  If new-onset atrial fibrillation occurred within this group, the rivaroxaban drug dose was increased from 10mg once-daily to 20mg once-daily (or 15mg once-daily in patients with moderate renal dysfunction as per drug label) plus acetylsalicyclic acid 75mg to 100mg once-daily; acetylsalicyclic acid was discontinued at three months post-TAVR.
Period: Overall Study
Arm/Group | ASA + Clopidogrel | Rivaroxaban + ASA
Started | 116 | 115
Completed | 101 | 97
Not Completed | 15 | 18
Not completed — Death | 2 | 3
Not completed — were not scanned | 8 | 13
Not completed — scans could not be evaluated | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASA + Clopidogrel | Rivaroxaban + ASA | Total
Number analyzed (Participants) | 116 | 115 | 231
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.5 (6.2) | 79.7 (7.3) | 80.1 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 41 | 83
  Male | 74 | 74 | 148
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body-mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.8 (5.1) | 27.7 (6.5) | 27.8 (5.8)
Hypertension [Count of Participants; unit: Participants] | 95 | 98 | 193
Diabetes Mellitus [Count of Participants; unit: Participants] | 27 | 21 | 48
STS risk score [Mean (Standard Deviation); unit: %] | 3.0 (2.1) | 2.8 (1.5) | 2.9 (1.8)
STS risk category - High [Count of Participants; unit: Participants] — The risk model of the Society of Thoracic Surgeons (STS) uses an algorithm that is based on the presence of coexisting illnesses to predict 30-day operative mortality. The STS score equals the predicted mortality expressed as a percentage.
  A score of greater than 8% indicates high risk, 3 to 8% intermediate risk, and les than 3% low risk.
  Participants | 3 | 1 | 4
STS risk category - Intemediate [Count of Participants; unit: Participants] — The risk model of the Society of Thoracic Surgeons (STS) uses an algorithm that is based on the presence of coexisting illnesses to predict 30-day operative mortality. The STS score equals the predicted mortality expressed as a percentage.
  A score of greater than 8% indicates high risk, 3 to 8% intermediate risk, and les than 3% low risk.
  Participants | 35 | 37 | 72
STS risk category - low [Count of Participants; unit: Participants] — The risk model of the Society of Thoracic Surgeons (STS) uses an algorithm that is based on the presence of coexisting illnesses to predict 30-day operative mortality. The STS score equals the predicted mortality expressed as a percentage.
  A score of greater than 8% indicates high risk, 3 to 8% intermediate risk, and les than 3% low risk.
  Participants | 78 | 77 | 155
Congestive Heart Failure [Count of Participants; unit: Participants] | 52 | 52 | 104
Coronary Artery Disease [Count of Participants; unit: Participants] | 36 | 42 | 78
Previous stroke [Count of Participants; unit: Participants] | 6 | 11 | 17
Peripheral Artery disease [Count of Participants; unit: Participants] | 10 | 10 | 20
Previous venous thromboembolism [Count of Participants; unit: Participants] | 1 | 1 | 2
Permanent Pacemaker [Count of Participants; unit: Participants] | 14 | 14 | 28
Chronic obstructive pulmonary disease [Count of Participants; unit: Participants] | 16 | 19 | 35
Glomerular filtration rate [Mean (Standard Deviation); unit: ml/min/1.73m2] | 76.6 (19.4) | 73.6 (19.2) | 75.1 (19.3)
Valve type - balloon-expandable [Count of Participants; unit: Participants] | 54 | 52 | 106
Valve type - Self-expandable [Count of Participants; unit: Participants] | 62 | 63 | 125
Valve type - Supra-annular leaflet position [Count of Participants; unit: Participants] | 46 | 37 | 83
Valve-in-valve [Count of Participants; unit: Participants] | 1 | 3 | 4
Post TAVR Echo - Aortic-valve-area [Mean (Standard Deviation); unit: cm2] | 1.8 (0.5) | 1.8 (0.5) | 1.8 (0.5)
Post TAVR Echo - mean aortic-valve gradient [Mean (Standard Deviation); unit: mm Hg] | 11 (4) | 11 (5) | 11 (4)
Post TAVR Echo - Left Ventricular ejection fraction [Mean (Standard Deviation); unit: %] | 56 (10) | 55 (11) | 56 (11)
Paravalvular aortic regurgitation - none or trace [Count of Participants; unit: Participants] | 96 | 94 | 190
Paravalvular aortic regurgitation - Mild [Count of Participants; unit: Participants] | 19 | 19 | 38
Paravalvular aortic regurgitation - moderate or severe [Count of Participants; unit: Participants] | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Rate of Patients With at Least One Prosthetic Leaflet With >50% Motion Reduction as Assessed by Cardiac 4DCT-scan
Description: Reduced systolic leaflet excursion is classified as: (I) normal, (II) mildly reduced (<50%), (III) moderate to severely reduced (>50%), and (IV) immobile. Reduced systolic leaflet excursion is considered significant when it is > 50% or immobile. Quantitative assessment of leaflet motion is performed with a blood pool inversion volume rendered cine reconstruction throughout the cardiac cycle evaluating the bioprosthetic leaflets.
Time Frame: 3 months
Population: Intention-to-treat (ITT) study population
Measure: Count of Participants; unit: Participants
Arm/Group | ASA + Clopidogrel | Rivaroxaban + ASA
Number analyzed (Participants) | 101 | 97
Participants | 11 | 2
Statistical Analysis 1: Comparison: ASA + Clopidogrel vs Rivaroxaban + ASA; Test type: Superiority; p = 0.01, Fisher Exact; The Fisher's exact probability test was used to compare the percentages of patients with the primary end point between the treatment groups

2. Secondary Outcome: The Rate of Prosthetic Leaflets With > 50% Motion Reduction as Assessed by Cardiac 4DCT-scan
Description: The rate of prosthetic leaflets with RLM> grade 3 as assessed by cardiac 4DCT
Time Frame: 3 months
Population: Intention-to-treat (ITT) study population
Measure: Number; unit: leaflets
Units Other Than Participants: leaflets
Arm/Group | ASA + Clopidogrel | Rivaroxaban + ASA
Number analyzed (Participants) | 101 | 97
Number analyzed (leaflets) | 303 | 291
leaflets | 14 | 3

3. Secondary Outcome: The Rate of Patients With at Least One Prosthetic Leaflet With Thickening as Assessed by Cardiac 4DCT-scan
Description: The rate of patients with at least one prosthetic leaflet with hypoattenuated leaflet thickening (HALT) as assessed by cardiac 4DCT.
Time Frame: 3 months
Population: Intention-to-treat (ITT) study population
Measure: Count of Participants; unit: Participants
Arm/Group | ASA + Clopidogrel | Rivaroxaban + ASA
Number analyzed (Participants) | 102 | 97
Participants | 33 | 12

4. Secondary Outcome: The Rate of Prosthetic Leaflets With Thickening as Assessed by Cardiac 4DCT-scan
Description: The rate of prosthetic leaflet with HALT as assessed by cardiac 4DCT-scan
Time Frame: 3 months
Population: Intention-to-treat (ITT) study population
Measure: Number; unit: Leaflets
Units Other Than Participants: Leaflets
Arm/Group | ASA + Clopidogrel | Rivaroxaban + ASA
Number analyzed (Participants) | 102 | 97
Number analyzed (Leaflets) | 306 | 291
Leaflets | 53 | 16

5. Secondary Outcome: Aortic Transvalvular Mean Pressure Gradient (mmHg) as Determined by Transthoracic Echocardiography.
Description: Transprosthetic mean pressure gradiënt as determined by transthoracic echocardiography at three months after randomization.
  scale [0-100]
Time Frame: 3 months
Population: Intention-to-treat (ITT) study population
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | ASA + Clopidogrel | Rivaroxaban + ASA
Number analyzed (Participants) | 105 | 102
mm Hg | 10 (5) | 10 (5)
Statistical Analysis 1: Comparison: ASA + Clopidogrel vs Rivaroxaban + ASA; Test type: Superiority; p = 0.01, Fisher Exact

6. Secondary Outcome: Effective Orifice Area (cm^2) as Determined by Transthoracic Echocardiography.
Description: Effective orifice area (cm2) as determined by transthoracic echocardiography at three months after randomization.
  scale [0.1-4.0]
Time Frame: 3 months
Population: Intention-to-treat (ITT) study population
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | ASA + Clopidogrel | Rivaroxaban + ASA
Number analyzed (Participants) | 105 | 102
cm2 | 1.8 (0.4) | 1.8 (0.5)

7. Secondary Outcome: Death Assessed in the Main GALILEO Study and Analyzed in the GALILEO-4D Substudy With Regards to Occurence of the Leaflet Abnormalities (HALT) - as Exploratory Analysis.
Description: Death, Dichotomization by HALT
Time Frame: 3 months
Population: Intention-to-treat (ITT) study population, subgroup of patients with analysable scans
Measure: Count of Participants; unit: Participants
Groups:
- HALT (-): Hypoattenuated leaflet thickening (-)
- HALT (+): Hypoattenuated leaflet thickening (+)
Arm/Group | HALT (-) | HALT (+)
Number analyzed (Participants) | 151 | 44
Participants | 0 | 0

8. Secondary Outcome: Death Assessed in the Main GALILEO Study and Analyzed in the GALILEO-4D Substudy With Regards to Occurence of the Leaflet Abnormalities (RLM)- as Exploratory Analysis.
Description: Death, Dichotomization by RLM
Time Frame: 3 months
Population: Intention-to-treat (ITT) study population, subgroup of patients with analysable scans
Measure: Count of Participants; unit: Participants
Groups:
- RLM>2 (-): Reduced Leaflet Motion >2 (-)
- RLM(+): Reduced Leaflet Motion >2 (+)
Arm/Group | RLM>2 (-) | RLM(+)
Number analyzed (Participants) | 169 | 25
Participants | 0 | 0

9. Secondary Outcome: Thromboembolic Event Assessed in the Main GALILEO Study and Analyzed in the GALILEO-4D Substudy With Regards to Occurence of the Leaflet Abnormalities (HALT)- as Exploratory Analysis.
Description: Thromboembolic event, Dichotomization by HALT
Time Frame: 3 months
Population: Intention-to-treat (ITT) study population, subgroup of patients with analysable scans
Measure: Count of Participants; unit: Participants
Arm/Group | HALT (-) | HALT (+)
Number analyzed (Participants) | 151 | 44
Participants | 2 | 0

10. Secondary Outcome: Thromboembolic Event Assessed in the Main GALILEO Study and Analyzed in the GALILEO-4D Substudy With Regards to Occurence of the Leaflet Abnormalities (RLM) - as Exploratory Analysis.
Description: Thromboembolic event, Dichotomization by RLM
Time Frame: 3 months
Population: Intention-to-treat (ITT) study population, subgroup of patients with analysable scans
Measure: Count of Participants; unit: Participants
Arm/Group | RLM>2 (-) | RLM(+)
Number analyzed (Participants) | 169 | 25
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: 90 days
Description: Adverse event reporting was captured via the Main Galileo trial (Global Study Comparing a rivAroxaban-based Antithrombotic Strategy to an antipLatelet-based Strategy After Transcatheter aortIc vaLve rEplacement to Optimize Clinical Outcomes) NCT02556203
Arm/Group | ASA + Clopidogrel | Rivaroxaban + ASA
All-Cause Mortality (participants affected / at risk) | 2/116 | 3/115
Serious Adverse Events (participants affected / at risk) | 3/116 | 7/115
Other Adverse Events (participants affected / at risk) | 17/116 | 16/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASA + Clopidogrel (N=116) | Rivaroxaban + ASA (N=115)
Major bleeding event (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Thromboembolic event (Cardiac disorders) | 2 (2) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASA + Clopidogrel (N=116) | Rivaroxaban + ASA (N=115)
minor bleeding (Blood and lymphatic system disorders) | 17 (17) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-29): https://cdn.clinicaltrials.gov/large-docs/48/NCT02833948/Prot_SAP_000.pdf